CLINICAL TRIAL: NCT02421211
Title: A Phase 2, 2-panel, Open-label Randomized Study in Hepatitis C Virus Infected Subjects to Investigate the Pharmacokinetic Interactions Between Simeprevir and Ledipasvir in a Treatment Regimen Consisting of Simeprevir, Sofosbuvir and Ledipasvir in Treatment-naive Participants.
Brief Title: A Study to Investigate the Pharmacokinetic Interactions Between Simeprevir and Ledipasvir in a Treatment Regimen Consisting of Simeprevir, Sofosbuvir, and Ledipasvir in Treatment-naive Participants With Chronic Hepatitis C Virus Genotype 1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR106992; TMC435HPC2017 (Other: Janssen Sciences Ireland UC); 2015-000459-25 (EudraCT Number)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Simeprevir; Ledipasvir; Sofosbuvir
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Simeprevir; ledipasvir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panel 1 (Experimental): Participants will receive Simeprevir (SMV) 150 milligram (mg) capsule (Treatment A) along with Sofosbuvir (SOF) 400 mg tablet, orally, once daily (Treatment C) from Day 1 until Day 14 followed by SMV 150 mg capsule (Treatment A) along with fixed dose combination (FDC) tablet of 90 mg Ledipasvir (LDV)/400 mg SOF (Treatment B), orally, once daily from Day 15 until Day 70.
  Interventions: Drug: Simeprevir (SMV); Drug: Ledipasvir (LDV); Drug: Sofosbuvir (SOF)
- Panel 2 (Experimental): Participants will receive FDC tablet of 90 mg LDV/400 mg SOF (Treatment B), orally, once daily from Day 1 until Day 14 followed by SMV 150 mg capsule (Treatment A) along with FDC tablet of 90 mg LDV/400 mg SOF (Treatment B), orally, once daily from Day 15 until Day 56.
  Interventions: Drug: Simeprevir (SMV); Drug: Ledipasvir (LDV); Drug: Sofosbuvir (SOF)

INTERVENTIONS:
Drug: Simeprevir (SMV) — Participants will receive 150 milligram (mg) of SMV (Treatment A) once daily in Panel 1 and Panel 2.
Drug: Ledipasvir (LDV) — Participants will receive 90 mg of LDV once daily as FDC tablet with SOF (Treatment B) in Panel 1 and Panel 2.
Drug: Sofosbuvir (SOF) — Participants will receive 400 mg of SOF alone (Treatment C) in Panel 1 and as FDC tablet with LDV (Treatment B) once daily in Panel 2.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic interactions between simeprevir and ledipasvir in a treatment regimen consisting of simeprevir (SMV), sofosbuvir (SOF), and ledipasvir (LDV) in treatment-naive participants with chronic hepatitis C virus (HCV) genotype 1 infection.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), 2-panel, Phase 2, randomized (study medication assigned to participants by chance) study. The study will consist of 3 study phases: Screening Phase (5 weeks), an Open-label Treatment Phase (70 days for Panel 1 and 56 days for Panel 2), a Post-treatment Follow-up Phase (12 weeks after the actual end of treatment). Participants will receive a combination of the following treatments: Treatment A: SMV 150 milligram (mg) once daily; Treatment B: LDV 90 mg along with SOF 400 mg once daily; Treatment C: SOF 400 mg once daily. Participants will be randomly assigned to Panel 1 (Treatment AC followed by Treatment AB) and Panel 2 (Treatment B followed by Treatment AB). The total study duration will be approximately 27 weeks for participants in Panel 1 and 25 weeks for participants in Panel 2. Participants will be primarily accessed for pharmacokinetic parameters. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Body Mass Index (weight in kilogram [kg] divided by the square of height in meters) of 18.0 to 35.0 kilogram per square meter kg/m^2, extremes included
* Participants must be treatment-naive (that is, have not received prior treatment with any approved or investigational drug)
* Participants with HCV ribonucleic acid (RNA) plasma levels greater than (>) 10,000 international unit per milliliter (IU/ml) and lower than 6,000,000 international unit per milliliter (IU/ml) at screening
* Participants with absence of cirrhosis confirmed by FibroTest/Fibrosure score less or equal to 0.75 and an aspartate aminotransferase to platelet ration index less or equal to 2 or a Fibroscan less or equal to 14.6 kilopascale (kPA), performed within 6 months prior or during the screening period
* Participants with documented chronic HCV infection: diagnosis of HCV infection >6 months prior to screening, either by detectable HCV RNA, an HCV positive antibody test or presence of histological changes consistent with chronic hepatitis in a liver biopsy

Exclusion Criteria:

* Participant has infection/co-infection with HCV of a genotype other than genotype 1, human immunodeficiency virus (HIV) type 1 or 2
* Participant has any evidence of liver disease of non-HCV etiology. This includes, but is not limited to acute hepatitis A, active hepatitis B, drug- or alcohol-related liver disease, autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, non-alcoholic steatohepatitis, primary biliary cirrhosis, or any other non-HC liver disease considered clinically significant by the investigator
* Participant with significant co-morbidities, conditions or clinical significant findings during screening assessments that in the opinion of the investigator could compromise the participants' safety or could interfere with the Participant participating in and completing the study
* Participant received an organ transplant (other than cornea or hair transplant or skin graft)
* Participants have key protocol defined laboratory abnormalities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-05-19 (Actual); Primary Completion 2015-11-10 (Actual); Study Completion 2016-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (4):
- Belgium (4):
  - Antwerp
  - Brussels
  - Ghent
  - Leuven

REFERENCES:
- [Derived] Bourgeois S, Horsmans Y, Nevens F, van Vlierberghe H, Moreno C, Beumont M, Vijgen L, van Eygen V, Luo D, Hillewaert V, Van Remoortere P, van de Logt J, Ouwerkerk-Mahadevan S. Pharmacokinetic Interactions between Simeprevir and Ledipasvir in Treatment-Naive Hepatitis C Virus Genotype 1-Infected Patients without Cirrhosis Treated with a Simeprevir-Sofosbuvir-Ledipasvir Regimen. Antimicrob Agents Chemother. 2017 Nov 22;61(12):e01217-17. doi: 10.1128/AAC.01217-17. Print 2017 Dec. PMID 28971875

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 41 participants were enrolled in the study, among them 40 participants (20 per panel) were randomized and treated. One participant was early terminated from the study, due to withdrawal of consent before randomization to study drug. All randomized participants received study drug and were included in the intent to treat (ITT) population.
Groups:
- Panel 1:SMV 150mg(SOF 400mg[2weeks]+LDV 90/SOF 400mg[8 Weeks]): Participants received simeprevir (SMV) 150 milligram (mg) capsule and sofosbuvir (SOF) 400 mg tablet, orally, once daily from Day 1 until Day 14. From Day 15 until Day 70, participants received SMV 150 mg capsule and a fixed dose combination (FDC) tablet of 90 mg Ledipasvir (LDV)/400 mg SOF, orally and once daily.
- Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks): Participants received fixed dose combination (FDC) tablet of 90 mg LDV/400 mg SOF, orally, once daily from Day 1 until Day 14. From Day 15 until Day 56, participants received SMV 150 mg capsule and a FDC tablet of 90 mg LDV/400 mg SOF, orally and once daily.
Period: Overall Study
Arm/Group | Panel 1:SMV 150mg(SOF 400mg[2weeks]+LDV 90/SOF 400mg[8 Weeks]) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks)
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel 1:SMV 150mg(SOF 400mg[2weeks]+LDV 90/SOF 400mg[8 Weeks]) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Full Range); unit: years] | 50.5 [25 to 70] | 51 [26 to 62] | 51 [25 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Minimum Plasma Concentration (Cmin) of Simeprevir (SMV)
Description: The Cmin is the minimum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, and 24 hours post-dose on Day 14 and Day 28
Population: The ITT analysis set is defined as all participants who took at least 1 dose of SMV, LDV, or SOF.
Measure: Mean (Standard Deviation); unit: nanogram per Milliliters (ng/mL)
Groups:
- Panel 1: SMV 150 mg + SOF 400 mg (Day 14): Participants received simeprevir (SMV) 150 milligram (mg) capsule and sofosbuvir (SOF) 400 mg tablet, orally, once daily from Day 1 until Day 14.
- Panel 1: SMV 150mg+LDV 90mg/SOF 400mg (Day 28): From Day 15 until Day 70, participants received SMV 150 mg capsule and a fixed dose combination (FDC) tablet of 90 mg Ledipasvir (LDV)/400 mg SOF, orally and once daily.
Arm/Group | Panel 1: SMV 150 mg + SOF 400 mg (Day 14) | Panel 1: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 20
nanogram per Milliliters (ng/mL) | 2411 (3778) | 6701 (4179)
Statistical Analysis 1: Comparison: Panel 1: SMV 150 mg + SOF 400 mg (Day 14) vs Panel 1: SMV 150mg+LDV 90mg/SOF 400mg (Day 28); Test type: Superiority or Other; LS means ratio = 4.7, 90% CI 2-sided [3.4 to 6.5]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Simeprevir
Description: The Cmax is the maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, and 24 hours post-dose on Day 14 and Day 28
Population: The ITT analysis set is defined as all participants who took at least 1 dose of SMV, LDV, or SOF. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panel 1: SMV 150 mg + SOF 400 mg (Day 14) | Panel 1: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 19
ng/mL | 6767 (6362) | 13691 (7775)
Statistical Analysis 1: Comparison: Panel 1: SMV 150 mg + SOF 400 mg (Day 14) vs Panel 1: SMV 150mg+LDV 90mg/SOF 400mg (Day 28); Test type: Superiority or Other; LS means ratio = 2.3, 90% CI 2-sided [2.0 to 2.8]

3. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Simeprevir
Description: The AUCtau is the measure of the plasma drug concentration from time zero to end of dosing interval. It is used to characterize drug absorption.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, and 24 hours post-dose on Day 14 and Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram hour per Milliliters (ng*h/mL)
Arm/Group | Panel 1: SMV 150 mg + SOF 400 mg (Day 14) | Panel 1: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 19
nanogram hour per Milliliters (ng*h/mL) | 100492 (115868) | 243564 (159124)
Statistical Analysis 1: Comparison: Panel 1: SMV 150 mg + SOF 400 mg (Day 14) vs Panel 1: SMV 150mg+LDV 90mg/SOF 400mg (Day 28); Test type: Superiority or Other; LS means ratio = 3.1, 90% CI 2-sided [2.4 to 3.8]

4. Primary Outcome: Minimum Plasma Concentration (Cmin) of Ledipasvir (LDV)
Description: The Cmin is the minimum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, and 24 hours post-dose on Day 14 and Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Panel 2: LDV 90mg/SOF 400mg (Day 14): Participants received FDC tablet of 90 mg LDV/400 mg SOF, orally, once daily from Day 1 until Day 14.
- Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (Day 28): From Day 15 until Day 56, participants received SMV 150 mg capsule and a FDC tablet of 90 mg LDV/400 mg SOF, orally and once daily.
Arm/Group | Panel 2: LDV 90mg/SOF 400mg (Day 14) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 18
ng/mL | 319 (178) | 557 (307)
Statistical Analysis 1: Comparison: Panel 2: LDV 90mg/SOF 400mg (Day 14) vs Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (Day 28); Test type: Superiority or Other; LS means ratio = 1.7, 90% CI 2-sided [1.5 to 2.0]

5. Primary Outcome: Maximum Plasma Concentration (Cmax) of Ledipasvir
Description: The Cmax is the maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, and 24 hours post-dose on Day 14 and Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panel 2: LDV 90mg/SOF 400mg (Day 14) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 17
ng/mL | 556 (270) | 930 (466)
Statistical Analysis 1: Comparison: Panel 2: LDV 90mg/SOF 400mg (Day 14) vs Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (Day 28); Test type: Superiority or Other; LS means ratio = 1.6, 90% CI 2-sided [1.4 to 1.9]

6. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Ledipasvir
Description: AUCtau is defined as area under the analyte concentration versus time curve during dosing interval tau, calculated by linear-linear trapezoidal summation.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, and 24 hours post-dose on Day 14 and Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Panel 2: LDV 90mg/SOF 400mg (Day 14) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 17
ng*h/mL | 9868 (4930) | 17435 (8772)
Statistical Analysis 1: Comparison: Panel 2: LDV 90mg/SOF 400mg (Day 14) vs Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (Day 28); Test type: Superiority or Other; LS means ratio = 1.7, 90% CI 2-sided [1.6 to 2.0]

7. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Simeprevir
Description: The (Ctrough) is the plasma concentration before dosing or at the end of the dosing interval of any dose other than the first dose in a multiple dosing regimen.
Time Frame: Pre-dose on Day 14 and Day 28
Population: The Intent-to-treat (ITT) analysis set is defined as all participants who took at least 1 dose of SMV, LDV, or SOF. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per Milliliters (ng/mL)
Arm/Group | Panel 1: SMV 150 mg + SOF 400 mg (Day 14) | Panel 1: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 19 | 20
nanogram per Milliliters (ng/mL) | 3059 (4236) | 8453 (6455)

8. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Simeprevir
Description: The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, and 24 hours post-dose on Day 14 and Day 28
Population: as for outcome 2
Measure: Median (Full Range); unit: hour (H)
Arm/Group | Panel 1: SMV 150 mg + SOF 400 mg (Day 14) | Panel 1: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 19
hour (H) | 6.00 [4.00 to 12.00] | 6.00 [0.47 to 10.00]

9. Secondary Outcome: Average Plasma Concentration at Steady State (Cavg,ss) of Simeprevir
Description: The Cavg,ss is calculated as area under the plasma concentration-time curve during a dosing Interval (AUC[tau]) divided by the dosing interval (tau).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, and 24 hours post-dose on Day 14 and Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panel 1: SMV 150 mg + SOF 400 mg (Day 14) | Panel 1: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 19
ng/mL | 4196 (4833) | 10139 (6628)

10. Secondary Outcome: Fluctuation Index (FI) of Simeprevir
Description: Fluctuation index is defined as percentage fluctuation (variation between maximum and minimum concentration at steady state), calculated as: 100*([Cmax Cmin]/Cavg).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, and 24 hours post-dose on Day 14 and Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage fluctuation
Arm/Group | Panel 1: SMV 150 mg + SOF 400 mg (Day 14) | Panel 1: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 19
percentage fluctuation | 144 (55.5) | 84.4 (36.5)

11. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Ledipasvir
Description: as for outcome 7
Time Frame: Pre-dose on Day 14 and Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panel 2: LDV 90mg/SOF 400mg (Day 14) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 18
ng/mL | 376 (211) | 659 (406)

12. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Ledipasvir
Description: The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, and 24 hours post-dose on Day 14 and Day 28
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour
Arm/Group | Panel 2: LDV 90mg/SOF 400mg (Day 14) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 17
Hour | 4.07 [1.00 to 8.00] | 6.00 [3.93 to 10.00]

13. Secondary Outcome: Average Plasma Concentration at Steady State (Cavg,ss) of Ledipasvir
Description: as for outcome 9
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, and 24 hours post-dose on Day 14 and Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panel 2: LDV 90mg/SOF 400mg (Day 14) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 17
ng/mL | 411 (207) | 725 (364)

14. Secondary Outcome: Fluctuation Index (FI) of Ledipasvir
Description: as for outcome 10
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, and 24 hours post-dose on Day 14 and Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage fluctuation
Arm/Group | Panel 2: LDV 90mg/SOF 400mg (Day 14) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (Day 28)
Number analyzed (Participants) | 20 | 17
percentage fluctuation | 60.6 (19.7) | 51.2 (0.17)

15. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 10 Weeks for Panel 1 and 8 Weeks for Panel 2
Population: The ITT analysis set is defined as all participants who took at least 1 dose of SMV, LDV, or SOF.
Measure: Number; unit: number of participants
Groups:
- Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks): Participants received FDC tablet of 90 mg LDV/400 mg SOF, orally, once daily from Day 1 until Day 14. From Day 15 until Day 56, participants received SMV 150 mg capsule and a FDC tablet of 90 mg LDV/400 mg SOF, orally and once daily.
Arm/Group | Panel 1:SMV 150mg(SOF 400mg[2weeks]+LDV 90/SOF 400mg[8 Weeks]) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks)
Number analyzed (Participants) | 20 | 20
number of participants
  Adverse events | 17 | 15
  Serious adverse events | 2 | 0

16. Secondary Outcome: Percentage of Participants With On-treatment Virologic Response
Description: On-treatment virologic response was determined by hepatitis C virus (HCV) ribonucleic acid (RNA) results satisfying a specified threshold.
  The following thresholds were considered at any time point: less than (<) lower limit of quantification (LLOQ) undetectable, <LLOQ detectable and <LLOQ undetectable/detectable.
Time Frame: Week 1, up to EOT (Week 10 in Panel 1 and Week 8 in Panel 2)
Population: The ITT analysis set is defined as all participants who took at least 1 dose of SMV, LDV, or SOF.
Measure: Number; unit: percentage of participants
Arm/Group | Panel 1:SMV 150mg(SOF 400mg[2weeks]+LDV 90/SOF 400mg[8 Weeks]) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks)
Number analyzed (Participants) | 20 | 20
percentage of participants
  Week 1: >= 15 IU/mL | 65.0 | 60.0
  Week 1: < 15 IU/mL undetectable/detectable | 35.0 | 40.0
  Week 1: < 15 IU/mL detectable | 15.0 | 35.0
  Week 1: < 15 IU/mL undetectable | 20.0 | 5.0
  Week 2: >= 15 IU/mL | 25.0 | 35.0
  Week 2: < 15 IU/mL undetectable/detectable | 75.0 | 65.0
  Week 2: < 15 IU/mL detectable | 30.0 | 30.0
  Week 2: < 15 IU/mL undetectable (vRVR) | 45.0 | 35.0
  Week 4: >= 15 IU/mL | 0 | 5.0
  Week 4: < 15 IU/mL undetectable/detectable | 100.0 | 95.0
  Week 4: < 15 IU/mL detectable | 15.0 | 5.0
  Week 4: < 15 IU/mL undetectable (RVR) | 85.0 | 90.0
  Week 6: >= 15 IU/mL | 0 | 0
  Week 6: < 15 IU/mL undetectable/detectable | 100.0 | 100.0
  Week 6: < 15 IU/mL detectable | 0 | 5.0
  Week 6: < 15 IU/mL undetectable | 100.0 | 95.0
  Week 8: >= 15 IU/mL | 0 | 0
  Week 8: < 15 IU/mL undetectable/detectable | 100.0 | 100.0
  Week 8: < 15 IU/mL detectable | 0 | 0
  Week 8: < 15 IU/mL undetectable | 100.0 | 100.0
  Week 10: >= 15 IU/mL | 0 | NA — Week 10 is not applicable for Panel 2. The scheduled end of treatment visit for Panel 2 was Week 8.
  Week 10: < 15 IU/mL undetectable/detectable | 100.0 | NA — Week 10 is not applicable for Panel 2. The scheduled end of treatment visit for Panel 2 was Week 8.
  Week 10: < 15 IU/mL detectable | 0 | NA — Week 10 is not applicable for Panel 2. The scheduled end of treatment visit for Panel 2 was Week 8.
  Week 10: < 15 IU/mL undetectable | 100.0 | NA — Week 10 is not applicable for Panel 2. The scheduled end of treatment visit for Panel 2 was Week 8.

17. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 4 Weeks After the Actual EOT (SVR4) and 12 Weeks After the Actual EOT (SVR12)
Description: SVR4 or SVR12 is defined as sustained virologic response 4 or 12 weeks after the actual EOT the participant has HCV RNA <LLOQ detectable or undetectable.
Time Frame: 4 weeks after EOT (Week 4 of follow-up phase in Panel 1 and Panel 2) and 12 weeks after EOT (Week 12 of follow-up phase in Panel 1 and Panel 2)
Population: The ITT analysis set is defined as all participants who took at least 1 dose of SMV, LDV, or SOF.
Measure: Number; unit: percentage of participants
Arm/Group | Panel 1:SMV 150mg(SOF 400mg[2weeks]+LDV 90/SOF 400mg[8 Weeks]) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks)
Number analyzed (Participants) | 20 | 20
percentage of participants
  SVR4 | 100 | 100
  SVR12 | 100 | 100

18. Secondary Outcome: Percentage of Participants With On-treatment Failure
Description: On-treatment failure is defined as participants who did not achieve SVR12 and with confirmed detectable HCV RNA at the actual end of treatment. This was to include participants with: 1) Viral breakthrough, defined as a confirmed increase of greater than (>)1 log10 in HCV RNA from nadir, or confirmed HCV RNA of >100 IU/mL in participants whose HCV RNA had previously been <LLOQ while on treatment; 2) Other with confirmed detectable HCV RNA at the actual end of treatment (example, completed, discontinued due to AEs, withdrawal of consent).
Time Frame: Day 70 in Panel 1 and Day 56 in Panel 2
Population: The ITT analysis set is defined as all participants who took at least 1 dose of SMV, LDV, or SOF.
Measure: Number; unit: percentage of participants
Arm/Group | Panel 1:SMV 150mg(SOF 400mg[2weeks]+LDV 90/SOF 400mg[8 Weeks]) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks)
Number analyzed (Participants) | 20 | 20
percentage of participants | 0 | 0

19. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Participants who did not achieve SVR12, with undetectable HCV RNA at the actual end of study drug treatment and confirmed HCV RNA greater than or equal to (>=) LLOQ during follow-up.
Time Frame: Up to Week 12 follow-up phase after EOT
Population: The ITT analysis set is defined as all participants who took at least 1 dose of SMV, LDV, or SOF.
Measure: Number; unit: percentage of participants
Arm/Group | Panel 1:SMV 150mg(SOF 400mg[2weeks]+LDV 90/SOF 400mg[8 Weeks]) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks)
Number analyzed (Participants) | 20 | 20
percentage of participants | 0 | 0

20. Secondary Outcome: Number of Participants Not Achieving Sustained Virologic Response (SVR) Showing Emerging Mutation in HCV Nonstructural Protein 3/4A (NS3/4A), Nonstructural Protein 5A (NS5A), and Nonstructural Protein 5B (NS5B) Sequence
Time Frame: Up to end of follow-up phase (Week 12 of follow-up phase) in Panel 1 and Panel 2
Population: The ITT analysis set is defined as all participants who took at least 1 dose of SMV, LDV, or SOF. Since the data was to be analysed in the participants who did not achieve SVR, but all the participants achieved SVR in the study. Therefore the data was not collected for this outcome measure.
Arm/Group | Panel 1:SMV 150mg(SOF 400mg[2weeks]+LDV 90/SOF 400mg[8 Weeks]) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 10 Weeks for Panel 1 and 8 Weeks for Panel 2
Arm/Group | Panel 1:SMV 150mg(SOF 400mg[2weeks]+LDV 90/SOF 400mg[8 Weeks]) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks)
Serious Adverse Events (participants affected / at risk) | 2/20 | 0/20
Other Adverse Events (participants affected / at risk) | 17/20 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panel 1:SMV 150mg(SOF 400mg[2weeks]+LDV 90/SOF 400mg[8 Weeks]) (N=20) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks) (N=20)
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panel 1:SMV 150mg(SOF 400mg[2weeks]+LDV 90/SOF 400mg[8 Weeks]) (N=20) | Panel 2: SMV 150mg+LDV 90mg/SOF 400mg (8 Weeks) (N=20)
Vertigo (Ear and labyrinth disorders) | 0 | 1
Eye irritation (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 1
Catheter site paraesthesia (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Angular cheilitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Genital abscess (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 3
Paraesthesia (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Breast atrophy (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 11 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 2 | 1
Vasculitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.